CLINICAL TRIAL: NCT07028112
Title: Impact de la Surcharge en Fer Sur l'Incidence Des Complications hépatiques Chez Les Patients allogreffés de Cellules Souches hématopoïétiques à Plus de 10 Ans de la Greffe
Brief Title: Impact of Iron Overload on the Incidence of Liver Complications in Long-Term Survivors (≥10 Years) of Allogeneic Hematopoietic Stem-Cell Transplantation.
Acronym: AlloFer
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH250402
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Iron Overload; Hemosiderosis; Liver Diseases; Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: Iron overload; Liver fibrosis; Elastography; Long-term complications; Allogeneic hematopoietic stem-cell transplantation; graft-versus-host disease
MeSH Terms: conditions — Iron Overload; Hemosiderosis; Liver Diseases; Liver Cirrhosis; Graft vs Host Disease | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Additional blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AlloFer cohort: Adults transplanted at Hôpital Saint Louis (2004-2014) and alive ≥10 years post allo HSCT; evaluated once during routine annual follow up
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Participants undergo one routine visit blood draw and non invasive liver stiffness measurement. Retrospective data are abstracted from medical records.

SUMMARY:
This single-center, non interventional cohort study investigates whether chronic iron overload influences the incidence of liver complications in adults who are at least 10 years beyond allogeneic hematopoietic stem cell transplantation (allo HSCT). Approximately 400-500 survivors transplanted at Hôpital Saint Louis between January 2004 and December 2014 will be evaluated. Transplant characteristics, prior iron overload therapy, and historical hepatic events will be collected through the Promise database. At the same time, the prospective visit will include laboratory panels and non invasive liver stiffness measurement by FibroScan or shear wave elastography. The study's primary objective is to assess the impact of iron overload on the incidence of hepatic complications in patients more than 10 years after an allogeneic hematopoietic stem cell transplantation. Secondary aims include describing the spectrum and frequency of hepatic complications, determining risk factors (including graft versus host disease, conditioning regimen, and comorbidities), and evaluating the long term effectiveness of previous iron reduction treatments (phlebotomy or chelation). Results will clarify whether monitoring and treating iron overload in long term allo HSCT survivors can prevent late hepatic morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at enrollment
* Allogeneic HSCT performed at Hôpital Saint Louis between 2004/01/01 and 2014/12/31
* Alive and attending routine annual follow up within the two years of the study
* Having given his non-opposition to study after understand overall aims
* With health insurance coverage
* Follow up consultation at Saint-Louis Hospital

Exclusion Criteria:

* Patient under legal protection (protection of the court, or in curatorship or guardianship).

not in relapse of the hematological disease at the time of inclusion.

• Patients under 45 Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) who received allo HSCT at Hôpital Saint Louis (2004/01/01 and 2014/12/31) and are alive and attending annual follow up ≥10 years post transplant.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | Up to 24 months
  From any hepatic complication ≥ 10 years after allogeneic HSCT

SECONDARY OUTCOMES:
Overall free survival of any hepatic complication ≥ 10 years after HSCT | Up to 24 months
  Survival without hepatic complication
Event free survival from liver fibrosis ≥ 10 years after HSCT | Up to 24 months
  Time from HSCT to first diagnosis of liver fibrosis by elastography (FibroScan® ≥ 8 kPa or shear wave ≥ 7 kPa).
  baseline to fibrosis diagnosis
Event free survival for each specific hepatic complication ≥ 10 years after HSCT | Up to 24 months
  Separate analyses for cirrhosis, portal hypertension, hepatic GVHD, viral hepatitis, steatosis, etc
Event free survival from iron overload ≥ 10 years after HSCT | Up to 24 months
  Time from HSCT to first diagnosis of iron overload
Efficacy of curative treatments for iron overload in preventing hepatic complications | Up to 24 months
  International non-proprietary names, dates and doses of treatments received for iron overload ≥ 10 years after HSCT

IPD SHARING:
Plan to Share IPD: Undecided